CLINICAL TRIAL: NCT02533258
Title: POST-MARKETING SURVEILLANCE STUDY TO OBSERVE INLYTA (REGISTERED) TREATMENT DOSING PATTERN, SAFETY AND EFFECTIVENESS IN TAIWAN REAL WORLD ROUTINE PRACTICE
Brief Title: Post-Marketing Surveillance Study To Observe INLYTA® Treatment Dosing Pattern, Safety And Effectiveness In Taiwan Real World Routine Practice
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A4061076; NCT02533258 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2015-08-24; First posted 2015-08-26 (Estimated); Results first posted 2017-10-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Renal Cell Carcinoma
Keywords: advanced renal cell carcinoma, disease progression, sunitinib, interferon alpha
MeSH Terms: conditions — Carcinoma, Renal Cell; Disease Progression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a post-marketing Surveillance study to observe INLYTA® treatment dosing pattern, safety and effectiveness in Taiwan real world routine practice. The primary objective of this registry is to monitor the dose adjustment of INLYTA® in real world routine practice. The secondary objectives include safety profile, objective response rate, and progression-free rate in real world routine practice.

DETAILED DESCRIPTION:
This is a multi-center chart review registry on mRCC patients treated with axitinib. Primary objective is the dose adjustment. Secondary objectives are safety profile, objective response rate and progression free survival. Efficacy assessment will be based on investigators' judgment. Patients treated with 1st dose of axitinib between May 7, 2013 and June 30, 2015 will be enrolled. The follow-up time is 12 months. Prior therapies should include sunitinib or interferon alpha.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as advanced RCC by histology or cytology
* Patients using axitinib as therapy after failure of sunitinib or cytokine
* Patients received axitinib treatment and follow up in the health care center participating present registry
* Patients agree to participate and signed inform consent or IRB waiving of signed informed consent document is available

Exclusion Criteria:

* Patients with first dose of axitinib earlier than 7th May 2013
* Patients with first dose of axitinib later than 30th June 2015.
* Patients participating in clinical research involving axitinib
* Patients with hypersensitivity to axitinib or to any other component of axitinib
* Patients under 18-year of age
* Pregnant women.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: advanced renal cell carinoma with disease progression on sunitinib or interferon
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2016-05-12 (Actual); Study Completion 2016-05-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4061076&StudyName=Post-marketing%20Surveillance%20Study%20To%20Observe%20Inlyta%20%28registered%29%20Treatment%20Dosing%20Pattern%2C%20Safety%20And%20Effectiveness%20In%20Taiwan%20Real%20World%20Routine%20Practice

RESULTS

PARTICIPANT FLOW:
Groups:
- Axitinib (INLYTA): Participants diagnosed with advanced renal cell carcinoma (RCC) and received axitinib therapy as per routine clinical practice according to the label-packaging-dosing (LPD) under the physician's prescription were observed for 40 months.
Period: Overall Study
Arm/Group | Axitinib (INLYTA)
Started | 13
Completed | 5
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Death | 2
Not completed — Other | 1
Not completed — Economic factor | 1
Not completed — Progression of pleural effusion | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: Safety population included all the enrolled participants who received at least one dose of the axitinib.
Groups:
- Axitinib (INLYTA): Participants diagnosed with advanced RCC and received axitinib therapy as per routine clinical practice according to the LPD under the physician's prescription were observed for 40 months.
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Duration of Axitinib Treatment
Time Frame: From initiation of axitinib treatment up to the end of the study (up to 40 months)
Population: Efficacy population included all the participants who were enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 13
months | 15.2 (13.32) [8.01 to 24.11]

2. Primary Outcome: Mean Daily Dose of Axitinib
Time Frame: From initiation of axitinib treatment up to the end of the study (up to 40 months)
Population: Efficacy population included all the participants who were enrolled in the study.
Measure: Mean (Standard Deviation); unit: milligram
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 13
milligram | 9.24 (3.31)

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as percentage of participants with confirmed complete response (CR) or partial response (PR) according to response evaluation criteria in solid tumors (RECIST) version 1.1. CR was defined as disappearance of all target, non-target lesions and all lymph nodes decreased to non-pathological in size (less than [<]10 millimeter [mm] short axis). PR was defined as at least 30 percent (%) decrease in sum of diameters of target lesions taking as reference the baseline sum, without progression of non-target lesions, no appearance of new lesions. Progression of disease (PD) was defined as greater than equal to (>=) 20% increase in sum of diameters of the target lesions taking as reference the smallest sum on study (this included the baseline sum if that was the smallest on study) or unequivocal progression in non-target lesions or appearance of 1 or more new lesions. Response evaluation was based on investigators' judgment.
Time Frame: From initiation of axitinib treatment until PD or death from any cause (up to 40 months)
Population: Efficacy population included all the participants who were enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 13
percentage of participants | 7.69

4. Secondary Outcome: Duration of Response
Description: Duration of response was defined as time from first documentation of objective tumor response (CR or PR), that was subsequently confirmed, to the first documentation of PD or to death due to any cause, whichever occurred first as per RECIST version 1.1. CR was defined as disappearance of all target, non-target lesions and all lymph nodes decreased to non-pathological in size (<10 mm short axis). PR was defined as at least 30% decrease in sum of diameters of target lesions taking as reference the baseline sum, without progression of non-target lesions, no appearance of new lesions. PD was defined as >=20% increase in sum of diameters of the target lesions taking as a reference smallest sum on study (this included the baseline sum if that was the smallest on study) or unequivocal progression in non-target lesions or appearance of 1 or more new lesions.
Time Frame: From initiation of axitinib treatment until PD or death from any cause (up to 40 months)
Population: Efficacy population included all the participants who were enrolled in the study. Here 'number of participants analyzed' signifies participants who achieved a confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 1
months | 1 [NA to NA] — Upper and lower limits of 95% confidence interval were not estimable since only 1 participant had event and analyzed for this outcome measure.

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined as the time duration in months from start of study treatment to the first documentation of PD or to death due to any cause, whichever occured first. PD was assessed by RECIST version 1.1. and defined as >=20% increase in the sum of the diameters of the target lesions taking as a reference the smallest sum on study (this included the baseline sum if that was the smallest on study) or unequivocal progression in non-target lesions or the appearance of 1 or more new lesions. Progression free survival based on investigators' judgment on medical records was calculated.
Time Frame: From initiation of axitinib treatment until PD or death from any cause (up to 40 months)
Population: Efficacy population included all the participants who were enrolled in the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 13
months | 32.73 [3.57 to NA] — The upper limit of 95% confidence interval was not reached at the time of data cut-off.

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life- threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. A treatment-emergent AE was defined as an event that emerged during the treatment period that was absent before treatment, or worsened during the treatment period relative to the pretreatment state. AEs included both serious and non--serious events.
Time Frame: From initiation of axitinib treatment up to end of the study (up to 40 months)
Population: Safety population included all the enrolled participants who received at least one dose of the axitinib.
Measure: Number; unit: participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 13
participants
  AEs | 11
  SAEs | 2

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) by Severity
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of the AEs was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Grade 1= mild; Grade 2= moderate; Grade 3= severe; Grade 4= life-threatening or disabling; Grade 5= death related to AE.
Time Frame: From initiation of axitinib treatment up to end of the study (up to 40 months)
Population: Safety population included all the enrolled participants who received at least one dose of the axitinib. Here 'number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 11
participants
  Grade 1 | 5
  Grade 2 | 3
  Grade 3 | 3
  Grade 4 | 0
  Grade 5 | 0

8. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (AEs)
Description: A treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug.
Time Frame: From initiation of axitinib treatment up to end of the study (up to 40 months)
Population: as for outcome 7
Measure: Number; unit: participants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 11
participants | 8

9. Secondary Outcome: Number of Participants Discontinued Due to Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship.
Time Frame: From initiation of axitinib treatment up to end of the study (up to 40 months)
Population: as for outcome 7
Measure: Number; unit: partcicipants
Arm/Group | Axitinib (INLYTA)
Number analyzed (Participants) | 11
partcicipants | 1

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Axitinib (INLYTA)
Serious Adverse Events (participants affected / at risk) | 2/13
Other Adverse Events (participants affected / at risk) | 10/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (INLYTA) (N=13)
Dissecting aortic aneurysm type B (Vascular disorders) | 1
Weight decreased (Investigations) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Oliguria (Renal and urinary disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 1
Anuria (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Axitinib (INLYTA) (N=13)
Hypertension (Vascular disorders) | 3
Fatigue (General disorders) | 2
Hepatotoxicity (Hepatobiliary disorders) | 1
Hernia (General disorders) | 1
Malaise (General disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Dry eye (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 3
Epigastric discomfort (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood lactate dehydrogenase increased (Investigations) | 1
Weight decreased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypophagia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Insomnia (Psychiatric disorders) | 2
Proteinuria (Renal and urinary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.